CLINICAL TRIAL: NCT06295978
Title: Prognostic Value of Cardiovascular Risk of sST2, suPAR and High-sensitivity Troponin I in Patients With Acute Chest Pain
Brief Title: Multimarker Approach in Acute Chest Pain
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Piccioni Andrea, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4896
Record Dates: First submitted 2023-02-15; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Disease Other
Keywords: Biomarkers; Chest pain; suPAR; sST2
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biochemical marker assays — DOSAGE BIOMARKERS

SUMMARY:
Chest pain is one of the most common causes of access in the Emergency Room, and it can be a clinical manifestation of a broad spectrum of diseases including those 'time dependent' conditions such as acute coronary syndrome (ACS). Diagnosis or exclusion of acute myocardial infarction (AMI) is a daily challenge in the emergency department (ED), especially when classic clinical criteria and ECG alone are unable to make the diagnosis. The ED physician has the extremely delicate task of managing patients with chest pain and being able to frame them correctly; therefore, he needs to make differential diagnosis since chest pain can be caused by non-cardiac vascular events but also extra-cardiovascular events, such as pulmonary, neurological, osteoarticular, gastrointestinal and psychological. Recently, the importance of inflammatory processes and endothelial damage in cardiovascular disease has been highlighted, and consequently the focus has been on new markers, in a "multimarker" approach in which the strengths of each are combined together to provide an optimal solution to a clinical problem.

The data suggest how a future integration of these biomarkers in the routine approach to the patient with acute chest pain in the ED might allow a better patient stratification and proper management, allowing the clinician to make an early safe discharge or a timely admission for those who deserve in-depth diagnostic-therapeutic investigation.

DETAILED DESCRIPTION:
BACKGROUND: Chest pain is one of the most common causes of access in the Emergency Room, and it can be a clinical manifestation of a broad spectrum of diseases including those 'time dependent' conditions such as acute coronary syndrome (ACS). Diagnosis or exclusion of acute myocardial infarction (AMI) is a daily challenge in the emergency department (ED), especially when classic clinical criteria and ECG alone are unable to make the diagnosis. The ED physician has the extremely delicate task of managing patients with chest pain and being able to frame them correctly; therefore, he needs to make differential diagnosis since chest pain can be caused by non-cardiac vascular events but also extra-cardiovascular events, such as pulmonary, neurological, osteoarticular, gastrointestinal and psychological. Recently, the importance of inflammatory processes and endothelial damage in cardiovascular disease has been highlighted, and consequently the focus has been on new markers, in a "multimarker" approach in which the strengths of each are combined together to provide an optimal solution to a clinical problem.

The role of the biomarker sST2 has been widely explored in heart failure, so much so that it was included in the AHA guidelines in 2013 and 2017. Recently, several studies are also proposing a role of sST2 in the prognostic stratification of patients with Acute Coronary Syndrome and ischaemic heart disease, in association with other biomarkers even proposing a possible therapeutic differentiation.

Furthermore, current studies have explored the role of the suPAR biomarker in cardiovascular disease. Indeed, its serum levels, closely correlated with immune and inflammatory activation, reveal it as a promising prognostic indicator. Although its non-cardiac-specific nature limits its diagnostic value for heart disease, its added value in identifying patients at risk of adverse cardiovascular events, morbidity and mortality when used in a multi-marker approach has been highlighted.

The combined use of sST2 and suPAR with high-sensitivity troponins, as opposed to contemporary troponins, exploring complementary aspects of myocardial damage, could be a promising strategy to identify those patients who, although with early rule-out after evaluation in the emergency room, present a higher risk of occurrence of distant cardiovascular events, thus deserving to be subjected to a customised diagnostic-instrumental procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Patients who came to the emergency department with chest pain of presumable cardiac origin and uncertain etiologic diagnosis
* ECG not diagnostic for ischemia
* cTnI ultra within limits

Exclusion Criteria:

* STEMI
* Sepsis and viral infections
* Patients with ECG abnormalities that make it uninterpretable for ischemic purposes
* Patients with previous coronary events
* History of heart failure
* Known diagnosis of cardiovascular disease, acute or chronic, including pericarditis, myocarditis
* Conditions involving increases in sST2 and suPAR unrelated to cardiac causes, especially acute/chronic inflammatory or fibrotic conditions (inflammatory bowel disease, neoplasms, moderate-to-severe pulmonary fibrosis, chronic hepatopathy; autoimmune diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients entering the emergency department with chest pain or other typical symptoms suspected of ACS will be included in the study if they are adults, not pregnant, and meet the predetermined inclusion criteria. Furthermore, patients who sign written informed consent to participate in the study and to the processing of personal data
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The predictive value of markers for the risk of cardiovascular events in chest pain | 2 years
  Evaluate the medium-long term (1 year) predictive value of the sST2, suPAR and IL6 biomarkers in patients attending the emergency department for acute non-STEMI chest pain

SECONDARY OUTCOMES:
Multimarker approach to improve cardiovascular risk stratification | 2 years
  A multimarker approach in combination with high-sensitivity troponin (hsTnI), improve cardiovascular risk stratification

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No